CLINICAL TRIAL: NCT05052385
Title: Multi-centre Retrospective Study to Describe the Use and Outcomes of ECP in Combination With New Treatment Protocols in Acute and Chronic GvHD
Brief Title: ECP Combination Study
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019000902
Record Dates: First submitted 2021-07-08; First posted 2021-09-22 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Steroid Refractory GVHD
Keywords: Steroid refractory GVHD; Extracorporeal photopheresis; Ibrutinib; Ruxolitinib; ECP
MeSH Terms: interventions — ruxolitinib; Photopheresis; ibrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (6):
- ECP only (aGVHD patients): Patients treated with ECP and other Standard Of Care treatments (SOC)
  Interventions: Device: Extracorporeal photopheresis
- ECP and Ruxolitinib (aGVHD patients): Patients treated with ECP and Ruxolitinib
  Interventions: Drug: Ruxolitinib; Device: Extracorporeal photopheresis
- Ruxolitinib only (aGVHD patients): Patients treated with Ruxolitinib and other Standard Of Care treatments (SOC)
  Interventions: Drug: Ruxolitinib
- ECP only (cGVHD patients): Patients treated with ECP and other Standard Of Care treatments (SOC)
  Interventions: Device: Extracorporeal photopheresis
- ECP and treatment combination (cGVHD patients): Patients treated with ECP and Ruxolitinib or Ibrutinib
  Interventions: Drug: Ruxolitinib; Device: Extracorporeal photopheresis; Drug: Ibrutinib
- Treatment combination only (cGVHD patients): Patients treated with Ibrutinib and/or Ruxolitinib and other Standard Of Care treatments (SOC)
  Interventions: Drug: Ruxolitinib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Ruxolitinib — As per treating physician's decision - non interventional study
  Groups: ECP and Ruxolitinib (aGVHD patients); ECP and treatment combination (cGVHD patients); Ruxolitinib only (aGVHD patients); Treatment combination only (cGVHD patients)
Device: Extracorporeal photopheresis — As per treating physician's decision - non interventional study
  Groups: ECP and Ruxolitinib (aGVHD patients); ECP and treatment combination (cGVHD patients); ECP only (aGVHD patients); ECP only (cGVHD patients)
Drug: Ibrutinib — As per treating physician's decision - non interventional study
  Groups: ECP and treatment combination (cGVHD patients); Treatment combination only (cGVHD patients)

SUMMARY:
Extracorporeal photopheresis (ECP) offers an alternative to standard immunosuppression and shows an immunomodulatory rather than an immunosuppressive effect, which is associated with less toxicities and side effects. Additionally ECP has been shown to allow tapering of steroids and immunosuppressant agents which should be a goal of GvHD therapy.

ECP has been used for the management of GvHD since first described in 1994 and as its use has continued over the decades. The treatment was incorporated into a number of guidelines as a second line therapy in steroid refractory or steroid dependent GvHD patients. As well as being used in addition and after steroids, it is also used in combination with CNI Inhibitors, MMF and other immunosuppressant agents.

However, despite the current widespread use of ECP in the treatment of patients with GvHD, clinical data from randomized studies is limited and small prospective and retrospective trials are the main evidence base .This is also the case for other commonly used immunosuppressant agents, which have been used in GvHD since ECP was introduced.

The systematic review concluded that ECP is an effective therapy for oral, skin, and liver SR-cGVHD, with modest activity in lung and gastrointestinal SR-cGVHD.

In the USA Ibrutinib is the only FDA approved agent for second line cGvHD therapy once steroid therapy has failed and Ruxolitinib had been approved in the USA for the treatment of steroid refractory GvHD.

While studies have shown the effectiveness and safety of ECP in GvHD treatment, there is limited data to show how it is being used in combination with the recently approved agents.

Using existing registry data targeting centres where the newer agents are being used and enhancing the capture of treatment data we believe we can undertake a larger scale study, which will include the new treatment protocols. The aim of the current study is to improve the evidence basis on the potential benefit of ECP use as treatment of GVHD.

DETAILED DESCRIPTION:
This is a Registry Based Study (RBS) designed to collect data on the treatment behaviour of acute and chronic GvHD after HSCT. The data collection will be based on the EBMT registry, which so far consists of two questionnaires (Forms A and B), mainly covering the primary disease diagnostics, the status before and at HSCT, the type of HSCT (donor status, preparative regimen etc) and the survival status. With a new questionnaire Form C, which will be similar in design as the current forms used in the registry, we aim at collecting more information and additional data on GvHD characteristics and treatment (schedule, combination, disease states) for both chronic and acute GvHD EBMT will work with the selected sites to facilitate the collection of additional data as specified in section 4.

The data collected will all be retrospective and include up to 3 years of data covering 2017 onwards, from onset of GvHD that has failed to respond to steroids with a minimum data follow up of 6 months for acute and 1 year for chronic. Centres will be asked to select patients that meet the inclusion criteria and fill in Form C retrospectively. The amount of additional data required will depend on whether the centre selected fills in the more detailed Form B or the more minimum data set in Form A.

Criteria for centre selection will be based on:

* Centres that have expressed a willingness to participate in the study through a feasibility questionnaire that was sent out prior to the study or via Email confirmation
* Centres who have responded through the feasibility questionnaire
* Centres where there is prior knowledge of use of both Ruxolitinib/Ibrutinib and ECP or have responded as such in the feasibility questionnaire

ELIGIBILITY:
Inclusion Criteria:

Acute GvHD Patients

1. Patients who develop acute SR-GvHD after first HSCT and there is a minimum of 6 months follow up data in the database
2. Patients who initiate treatment with ECP or Ruxolitinib within 60 days of onset of SR aGvHD
3. Grade: II-IV only at time of treatment initiation
4. Patients who are ≥ 18 years at time of treatment initiation

Chronic GvHD Patients

1. Patients who develop chronic SR-GvHD after first HSCT and there is with a minimum of 1 year follow up data in the database
2. Patients who initiate treatment with ECP or Ruxolitinib or Ibrutinib within I year of the onset of SR-cGvHD
3. Severity: moderate to severe only at time of treatment initiation
4. Patients who are ≥ 18 years at time of treatment initiation

Exclusion Criteria:

Acute GvHD

1. Patients on a clinical trial for GvHD for an interventional drug to treat GvHD in the retrospective period
2. Patient is pregnant or breastfeeding
3. Grade I at time of SR GvHD treatment initiation
4. Patients who receive ECP or new treatment as prophylaxis
5. Patients initiating ECP or new treatment later than 60 days from onset on SR-aGvHD
6. Patients < 18 years at time of treatment initiation

Chronic GvHD

1. Patients on a clinical trial for an interventional drug to treat GvHD in the retrospective period
2. Patient is pregnant or breastfeeding
3. Chronic GvHD : Severity mild at time of SR GvHD treatment initiation
4. Patients who receive ECP or new treatment as prophylaxis
5. Patients initiating ECP or new treatment after 1 year onset of SR-cGvHD
6. Patients < 18 years at time of treatment initiation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute GvHD patients with HSCT who have failed steroids and developed SR-GvHD and are treated with either ECP or/and Ruxolitinib.
  Patients with HSCT who have developed chronic GvHD and failed to respond to steroids (SR-cGvHD) and are treated with either ECP or/and Ruxolitinib or/and Ibrutinib.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 3 months
  Partial or Complete response according to NIH/Glucksberg classification) at 3 months for acute GvHD since start of targeted* treatment for SR-GvHD
Overall response rate (Partial or Complete response according to NIH/Glucksberg classification) at 6 months for chronic GvHD since start of targeted* treatment for SR-GvHD | 6 months

SECONDARY OUTCOMES:
Efficacy of ECP | up to one year
  Organ specific response
Safety of ECP | Up to one year
  Incidence of Complications and infections
Safety of ECP | Up to one year
  Steroid sparing effects (decrease of dose or percentage)
Efficacy of ECP | Up to one year
  overall survival (Percentage at a fixed time)
Efficacy of ECP | Up to one year
  Non Relapse Mortality
Efficacy of ECP | Up to one year
  Duration of response
Efficacy of ECP | Up to one year
  Failure-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Penack, MD, Principal Investigator — European Society for Blood and Marrow Transplantation
Locations (38):
- Belgium (2):
  - Antwerp University, Antwerp
  - University of Liège, Liège
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - CHRU Angers, Angers
  - CHU de Limoges, Limoges
  - Institut de Cancerologie Lucien Neuwirth, Saint-Etienne
- Germany (4):
  - Bonn University, Bonn
  - University Hospital Essen, Essen
  - Universitaetsmedizin Mannheim, Mannheim
  - Robert_Bosch_Krankenhaus, Stuttgart
- George Papanicolaou General Hospital, Thessaloniki, Greece
- Rambam Medical Center, Haifa, Israel
- Italy (7):
  - H SS. Antonio e Biagio, Alessandria
  - ASST Papa Giovanni XXIII, Bergamo
  - Istituto Clinico Humanitas, Milan
  - Ospedale Civile, Pescara
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Universita Cattolica S. Cuore, Roma
  - S. Bortolo Hospital, Vicenza
- Medical University of Gdansk, Gdansk, Poland
- Fundeni Clinical Institute, Bucharest, Romania
- First State Pavlov Medical University of St. Petersburg, Saint Petersburg, Russia
- Spain (7):
  - ICO-Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - ICO - Hospital Duran i Reynals, Barcelona
  - Hosp. Reina Sofia, Córdoba
  - Hospital Univ. Virgen de las Nieves, Granada
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skanes University Hospital, Lund
- Turkey (Türkiye) (2):
  - Baskent University Hospital, Adana
  - Gazi University Faculty of Medicine, Ankara
- United Kingdom (5):
  - University Hospital Birmingham NHS Trust, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Kings College Hospital, London
  - Christie NHS Trust Hospital, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No